CLINICAL TRIAL: NCT07123363
Title: Effect of Bitopertin on the Liver and on Levels of Protoporphyrin IX in Bile, Blood, Liver, and Stool in Patients With Erythropoietic Protoporphyria/X-linked Protoporphyria and Increased Liver Stiffness and/or Liver Enzymes at Baseline
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: department leadership decided not to proceed with study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00118441
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Protoporphyria
Keywords: Erythropoietic Protoporphyria; X-linked Protoporphyria; Bitopertin
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bitopertin (Experimental): bitopertin 60 mg per day
  Interventions: Drug: bitopertin

INTERVENTIONS:
Drug: bitopertin — bitopertin 60 mg will be taken once daily by mouth
  Other Names: DISC-1459

SUMMARY:
The primary goal of this study is to assess safety and tolerability of bitopertin in subjects with Erythropoietic Protoporphyria (EPP) or X-linked Protoporphyria (XLP) and evidence of compensated liver disease.

DETAILED DESCRIPTION:
This in an open-label, investigator-initiated study of bitopertin (60 mg/day) in selected and carefully monitored participants with Erythropoietic Protoporphyria (EPP) or X-linked Protoporphyria (XLP) who have increased liver stiffness and/or elevated liver enzymes at baseline.This study is designed to evaluate whether bitopertin is effective in reducing hepatic and biliary levels of protoporphyrin IX (PP), which over time, with chronic and ongoing bitopertin treatment, will ameliorate and forestall progression of PP hepatopathy, providing an additional major benefit and reason for its chronic use in patients with EPP/XLP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of EEP or XLP that has been biochemically and genetically verified prior diagnosis of EPP or XLP
* Age 18-75 years
* Increased liver stiffness at baseline, defined as stiffness measurement [E value] by: Fibroscan >7 kPa; MRE that is >3.0 kPa; Velacur/Sonicincyte that is >6.0 kPa; and/or elevated liver enzymes: serum ALT > 2 X upper limit of normal (ULN), but not greater than 5 X ULN and/or serum AP > 2 X ULN, but not greater than 5 X ULN
* INR < 1.4
* Compensated liver disease at baseline, defined as lack of clinically evident ascites, encephalopathy, hepatocellular carcinoma, clinically evident icterus or jaundice, peripheral edema.
* Willingness and ability to volunteer and provide informed consent for a long-term study that will include liver biopsies and collection of bile from the second portion of the duodenum, at baseline and at the end of study. In addition, follow-up visits will be planned every 26 weeks throughout the study, with plans for repeat routine/safety labs at each visit and for measures of liver stiffness and markers of hepatic status and fibrosis (Fib-4, APRI, ELF, Fibrotest) performed once every 6 months.

Exclusion Criteria:

* Chronic hepatitis B, C, D, or E;
* Human immunodeficiency (HIV) infection;
* Alcohol use > 14 units/week for men or > 7 units/week for women;
* Pregnancy or breast feeding among women;
* Any known active malignancy other than small and localized squamous or basal cell carcinoma of the skin;
* Advanced or decompensated heart, lung, kidney, liver, or neuro-psychiatric disease;
* History of diagnosed depression or suicidality;
* History of diagnosed substance abuse or poor impulse control;
* Any other conditions that, in the opinion of the Investigator, renders the individual unfit to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | Week 104
  Number of treatment emergent adverse events (TEAE). Adverse events that begin after the first administration of study drug, or existing adverse events that worsen after the first dose of study drug will be considered TEAEs.

SECONDARY OUTCOMES:
Percent Change in Protoporphyrin IX (PP) Serum Levels | baseline to month 12, month 12 to month 24
  To assess effects of bitopertin on levels of protoporphyrin IX (PP) and other porphyrins in the whole blood, plasma, and red blood cells
Number of Participants with Change in Histopathology | baseline to month 24
  To assess effects of bitopertin on hepatic histopathology the number of participants with change in histopathologic evidence will be tracked. Histopathology consists of histopathologic evidence of hepatic fibrosis, necroinflammation, fat, cholestasis, bile plugs, birefringent brown deposits in the liver, or other histopathology, as estimated by an experienced hepato-pathologist.
Percent Change in Protoporphyrin IX (PP) Bile Levels | baseline to month 24
  the percent change of Protoporphyrin IX (PP) in bile will be used to assess effects of bitopertin on PP levels
Percent Change in Protoporphyrin IX (PP) Liver Levels | baseline to month 12, baseline to month 24
  the percent change in Protoporphyrin IX (PP) in the liver will be measured by change in liver stiffness measured by vibration controlled elastography with use of dedicated instruments designed for this purpose (Fibroscan, Velocur)
Percent Change in Protoporphyrin IX (PP) Stool Levels | baseline to month 24
  the percent change in Protoporphyrin IX (PP) in stool will be used to assess effects of bitopertin on PP levels

OTHER OUTCOMES:
Patient Global Impression of Severity | baseline, week 26, week 52, week 78, week 104
  Three items with total score range 3-15. Higher score indicates higher level of erythropoietic protoporphyria severity
Patient Global Impression of Change | baseline, week 26, week 52, week 78, week 104
  Five items with total score range 5-25. Higher score indicates erythropoietic protoporphyria have gotten worse since start of the study.
Patient-Reported Outcomes Measurement Information System - Social Isolation | baseline, week 26, week 52, week 78, week 104
  Seven items with total score range 3-15. Higher score indicates poor quality of life.
Serum of Level of Bitopertin | baseline, week 26, week 52, week 78, week 104
  Trough concentrations of bitopertin will measured by using HPLC-mass spectroscopic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Bonkovsky, MD, Principal Investigator — Atrium Health Wake Forest Baptist

IPD SHARING:
Plan to Share IPD: No